CLINICAL TRIAL: NCT03136939
Title: Study of IGRP-specific T Cell in Peripheral Blood of Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-420
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- type 1 diabetes
  Interventions: Other: No intervention
- type 2 diabetes
  Interventions: Other: No intervention
- healthy people
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
10 type 1 diabetes, 10 type 2 diabetes and 10 healthy controls matched with age and sex were enrolled in our study and their periphera blood mononuclear cells (PBMC) were isolated. We implemented ELISPOT(Enzyme-linked Immunospot Assay) to detect the interferon-γ (IFN-γ）which secreted by IGRP-specific T cell. Results were compared between these groups.

ELIGIBILITY:
Inclusion Criteria:

* the criteria of type 1 and type 2 diabetes

Exclusion Criteria:

* no diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients of diabetes and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
the rate of positive reactivation against the IGRP epitopes | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, the First Affiliated Hospital to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
IPD be shared while request by email